CLINICAL TRIAL: NCT00818129
Title: A Phase I, Randomized, Double-Blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7295 Following Single and Multiple Ascending Oral Dose Administration in Healthy Male Japanese Subjects
Brief Title: Study to Investigate Safety, Tolerability and PK Following Single and Multiple Ascending Doses of AZD7295 in Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dereck Tait, Medical Science Director, Anti-Viral EPT, Arrow Therapeutic Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1820C00001
Record Dates: First submitted 2008-12-24; First posted 2009-01-07 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
Keywords: Phase I; Japan; Japanese; oral solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD7295
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7295 — ascending single doses (start dose 90 mg), oral solution and then multiple ascending dose (tbd based on single dose results), oral solution
  Arms: 1
Drug: Placebo — multiple ascending dose (tbd based on single dose results), oral solution
  Arms: 2

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of single and multiple oral doses of AZD7295 in healthy male Japanese subjects. This will be done by comparing the effect of AZD7295 to placebo. The study will aslo investigate the absorption, distribution and disappearance of AZD7295 in the body.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent
* Healthy male Japanese volunteers aged 20-55 years
* BMI between 18 and 27 kg/m2
* Have negative screens for HIV, hepatitis B and C viruses and syphilis

Exclusion Criteria:

* Use of prescribed medication within 2 weeks prior to the dose of study medication
* Participation in another study that included drug treatment within 16 weeks before the start of the present study.
* History or presence of gastrointestinal, hepatic or renal disease or a condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* History of severe food or drug allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged relevant by the investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2008-12; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
AE, safety laboratory test (haematology, clinical chemistry, urinalysis), 12-lead ECG, BP, pulse rate, body temperature | During the study

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax, tmax, AUC, AUC0-t, CL/F, Vss/F, t1/2 , Cmin, Rac, etc) | Frequent sampling until 72 hours after single administration in Single Dose Part and until 72 hours after last administration (6 days administration) in Multiple Dose Part

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Tsukamoto, MD, Principal Investigator — Kyushu Clinical Pharmacolgy Reasearch Clinic
Locations (1):
- Research Site, Fukuoka, Fukuoka, Japan